CLINICAL TRIAL: NCT07148492
Title: Antireflux Suture In Laparoscopic One Anastomsis Gastric Bypass Surgery, A Randomised Control Trial
Brief Title: Antireflux Suture In One Anastomsis Gastric Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Saeed Sarwar, Dr, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 528/DME/KMC
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Reflux Disease, Gastro-Esophageal; Vomiting, Postoperative
MeSH Terms: conditions — Gastroesophageal Reflux; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antireflux suture group (Experimental): This group consist of patients in whom antireflux suture is taken
  Interventions: Procedure: Antireflux suture
- No Antireflux suture (Experimental): This group consist of patients in whom no antireflux suture is taken
  Interventions: Procedure: No Antireflux suture

INTERVENTIONS:
Procedure: Antireflux suture — Antireflux suture will be taken in this intervention group
  Arms: Antireflux suture group
Procedure: No Antireflux suture — Antireflux suture will not be taken in this intervention group
  Arms: No Antireflux suture

SUMMARY:
To prevent refulx symptoms in a type of bariatric surgery, a suture is taken.there is no enough evidence in support of or against the suture. our study aims to compare the symptoms of patients in whom the suture is taken and in those in whom it is not.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing one anastomosis gastric bypass surgery

Exclusion Criteria:

* Non consenting individuals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reflux disease | 3 months and 6 months postoperatively
  The incidence of gastroesophageal reflux will be measured after surgery

SECONDARY OUTCOMES:
Postoperative vomiting | At 3 months and 6 months postoperatively
  Incidence of postoperative vomiting will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber teaching hospital, Peshawar, Khyberpukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patients privacy may be breached